CLINICAL TRIAL: NCT05523128
Title: A Non-randomized, Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability, Kinetics and Efficacy of a Single Intravenous Infusion of ZS802 in Hemophilia A Subjects With Endogenous FVIII ≤2%.
Brief Title: The Efficacy and Safety of ZS802 in Chinese Hemophilia A Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022031
Record Dates: First submitted 2022-07-25; First posted 2022-08-31 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Gene therapy; Adeno-associated virus
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: Hemophilia A patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZS802 (Experimental): Single intravenous (i.v.) infusion of ZS802 Intervention: Gene Therapy / Gene Transfer
  Interventions: Genetic: ZS802

INTERVENTIONS:
Genetic: ZS802 — A novel, bioengineered adeno-associated viral (AAV) vector carrying human factor VIII variant. The dose levels are as follows: 1. 2.0×10^13vg/kg; 2. 6.0×10^13vg/kg.

SUMMARY:
A non-randomized, open-label, dose-escalation study to evaluate the safety, tolerability, kinetics and efficacy of a single intravenous infusion of ZS802 in hemophilia A subjects with endogenous FVIII ≤2%.

DETAILED DESCRIPTION:
This study will seek to determine the safety, tolerability, kinetics and efficacy of a single IV infusion of ZS802.

Hemophilia A is a genetic bleeding disorder resulting in the lack of ability to produce blood-clotting factor VIII (FVIII). Individuals with hemophilia A suffer repeated bleeding events, which can cause chronic joint disease and sometimes leads to death due to the inability for blood to clot efficiently. The current treatment is intravenous infusion of FVIII protein products, either prophylactically or in response to bleeding. ZS802 is an adeno-associated viral (AAV) vector designed to drive expression of the human factor VIII (hFVIII) transgene and raise circulating levels of endogenous FVIII.

6 patients will be enrolled sequentially every 3 weeks or more between cohorts and administered with single infusion of ZS802. Dose escalation may occur based on the safety and FVIII activity on steady state. The dose levels are as follows: 1. 2.0×10^13vg/kg; 2. 6.0×10^13vg/kg. Subjects will provide informed consent and then undergo screening assessments up to 6-8weeks prior administration of ZS802. All subjects will undergo 52 weeks safety and efficacy observation.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥18 years and ≤65years of age;
2. Confirmed diagnosis of hemophilia A, and endogenous FVIII ≤2%:

   1. <1% (<1 IU/dL) endogenous FVIII activity levels as historically documented by a certified laboratory or screening data results; OR
   2. 1%-2% (1-2 IU/dL) endogenous FVIII activity levels and >10 bleeding events per year (in the last 52 weeks prior to screening); OR
   3. 1%-2% (1-2 IU/dL) endogenous FVIII activity levels and on prophylaxis;
3. Have had ≥150 prior exposure days (EDs) to any recombinant and/or plasma-derived FVIII protein products.
4. Agree to use reliable barrier contraception and prohibition of sperm donation until 52 weeks after the administration of ZS802.
5. Subjects voluntarily participate and are fully informed, fully understand the research and can comply with the requirements of the research protocol, are willing to complete the research as planned, and voluntarily cooperate with the provision of biological samples for testing.

Exclusion Criteria:

1. Hypersensitivity to any component of the study drug (including immunosuppressants) or a condition that can not use.
2. Inability to tolerate immunosuppressants or steroid drugs.
3. Have no measurable FVIII inhibitor as assessed by laboratory; or documented no prior history of FVIII inhibitor.
4. Who have a history or are currently suffering from any of the following serious clinical diseases:

   1. History of malignancy or current presence of any malignancy;
   2. Have active autoimmune disease;
   3. Severe heart disease, including angina pectoris, myocardial infarction, heart failure, clinically significant congenital heart disease, heart valve disease, arrhythmia and atrioventricular block, etc.;
   4. Have underlying liver disease or history of liver disease (such as portal hypertension, ascites, splenomegaly, esophageal varices, hepatic encephalopathy or hepatic fibrosis);
   5. Have active hepatitis B infection (HBsAg positive or HBV-DNA positive) or active hepatitis C infection (HCVAb positive), or are currently receiving hepatitis B or hepatitis C antiviral therapy;
   6. Have history of chronic infection or other chronic disease that the Investigator considers to constitute an unacceptable risk;
   7. Diabetes mellitus that is poorly controlled after drug treatment;
   8. Uncontrolled hypertension or hypotension;
5. laboratory values:

   1. Hemoglobin<110g/L;
   2. Platelets<100×10^9/L;
   3. AST, ALT, alkaline phosphatase>2×ULN;
   4. Total bilirubin>1.5×ULN;
   5. Creatinine>ULN;
   6. Albumin<LLN;
   7. HIV antibody positive or Treponema pallidum antibody positive.
6. Have AAV5 capsid neutralizing antibody titers >1:5.
7. Those who have received clinical trials of gene therapy before screening, or have used FVIII clinical trial drugs within 1 month, or participated in other drug/device clinical trials within 3 months, or plan to participate in other clinical trials during this study.
8. Those who have planned surgery within 52 weeks after the infusion.
9. Those who donated or lost more than 400 mL of blood within 3 months before screening.
10. Those with epilepsy, history of mental illness (such as schizophrenia, depression, mania or anxiety) or obvious mental disorder, incapacitated or incapacitated by other reasons.
11. Patients with a history of drug abuse or alcoholism.
12. Investigators believe that subjects have poor compliance or are expected to be less likely to complete follow-up.
13. There are clinically significant diseases or other reasons that the researcher and/or collaborators consider unsuitable to participate in this researcher.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Baseline up to Week 52
  An adverse event (AE) is any medical occurrence, the event will not relate to the treatment.
Number of participants with clinically significant change from baseline in vital signs | Baseline up to Week 52
  Vital signs will be obtained with participants in the seated position, after having sat calmly for at least 5 minutes. The clinical significance of vital signs will be determined at the investigator's discretion.
Number of participants with clinically significant change from baseline in physical examination findings | Baseline up to Week 52
  Findings will be considered to be clinically significant based on the investigator's decision.
Number of participants with clinical laboratory abnormalities | Baseline up to Week 52
  Findings were considered to be clinically significant based on the investigator's decision.

SECONDARY OUTCOMES:
Vector-derived FVIII:C Activity | Baseline up to Week 52
  Peak and steady-state vector-derived circulating FVIII activity levels, and changes of FVIII activity levels after treatment compared with baseline.
Vector-derived FVIII antigen levels | Baseline up to Week 52
  Peak and steady-state vector-derived circulating FVIII antigen levels, and changes of FVIII antigen levels after treatment compared with baseline.
Vector shedding of ZS802 | Baseline up to Week 52
  Blood, saliva, urine and semen will be collected to assess clearance of vector genomes.
Antibody against AAV capsid protein | Baseline up to Week 52
  Immune response against AAV capsid will be evaluated by measurement of the binding antibody and neutralizing antibody against AAV capsid protein in plasma samples.

OTHER OUTCOMES:
Annualized bleeding rate changes from baseline | Baseline up to Week 52
  The number of bleeding episodes per participant will be recorded, and the annualized number of bleeding episodes was calculated.
Annualized FVIII consumption changes from baseline | Baseline up to Week 52
  The use of on-demand FVIII replacement therapy will be recorded by dose (IU/kg) administered, and the annualized use of FVIII replacement therapy will be calculated.
Number of target joints | Baseline up to Week 52
  The target joint is a minimum of three bleeds into a single joint within a consecutive 6-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when ZS802 is fully approved.
Supporting Information: Study Protocol
Time Frame: IPD will be shared with other researchers when ZS802 is fully approved.
Access Criteria: IPD will be shared with other researchers when ZS802 is fully approved.